CLINICAL TRIAL: NCT00738114
Title: Type 2 Diabetes in the Perioperative Period: Prevalence and Clinical Outcome
Brief Title: Diabetes in the Perioperative Period
Status: Completed | Type: Observational
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Guillermo Umpierrez, Principal Investigator, Emory University
Other Study IDs: IRB00011938
Record Dates: First submitted 2008-08-19; First posted 2008-08-20 (Estimated); Last update posted 2013-11-21 (Estimated); Status verified 2013-11

CONDITIONS: Hyperglycemia; Diabetes
Keywords: non-cardiac; surgery; mortality; morbidity; perioperative; period
MeSH Terms: conditions — Hyperglycemia; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: group without hyperglycemia (fasting blood glucose below 126mg/dl) approximately 1000 patients
- 2: group with hyperglycemia (fasting blood glucose above 125 mg/dl) or history of diabetes approximately 500 patients

SUMMARY:
High blood glucose levels in surgical patients with and without diabetes are associated with increased risk of medical complications and death. Over the short-term, high blood glucose can adversely affect fluid balance, impair immunologic response to infection, and promote inflammation and endothelial dysfunction (blood vessel function). Blood glucose control with intensive insulin therapy in patients with critical illness (very sick patients in intensive care unit) reduces the risk of multiorgan failure and systemic infections, and decreases short- and long-term mortality. High blood glucose has also been associated with poor outcome in non-critically ill patients admitted to general surgical and medical wards; however, intensive glycemic control is not aggressively pursued because of fear of hypoglycemia. A computerized search of biomedical journal literature from MEDLINE, PubMed, and Ovid from 1966 to 2008 provided very little information on the prevalence and outcome of high blood glucose during the perioperative period (before and after surgery) in non-critically ill patients. Therefore, the present study aims to evaluate the impact of high blood glucose, in large number of subjects with and without diabetes, during general (non-cardiac) surgery.

DETAILED DESCRIPTION:
We will perform a retrospective chart review of all patients who underwent non-cardiac surgery from 01/01/07 to 06/30/07 at Emory University Hospital as inpatient.

ELIGIBILITY:
Inclusion Criteria:

* patient undergoing non-cardiac surgery (inpatient only)

Exclusion Criteria:

* outpatient procedures, cardiac surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: all patients admitted for non-cardiac surgery during the period of 01/01/07 and 06/30/2007
Sampling Method: Probability Sample
Enrollment: 3184 (Actual)
Dates: Start 2008-08; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
assess impact of hyperglycemia and diabetes during the periop period on clinical outcome(mortality and morbidity)in patients undergoing general and non-cardiac surgery. | 01/01/07 - 06/30/2007

SECONDARY OUTCOMES:
determine the scope of clinical inertia in patients with diabetes and untreated hyperglycemia in patients undergoing non-cardiac surgery | 01/01/07 - 06/30/2007

CONTACTS AND LOCATIONS:
Overall Officials: Guillermo Umpierrez, MD, Principal Investigator — Emory University
Locations (1):
- Emory Universiy Hospital, Atlanta, Georgia, United States

REFERENCES:
- [Result] Frisch A, Chandra P, Smiley D, Peng L, Rizzo M, Gatcliffe C, Hudson M, Mendoza J, Johnson R, Lin E, Umpierrez GE. Prevalence and clinical outcome of hyperglycemia in the perioperative period in noncardiac surgery. Diabetes Care. 2010 Aug;33(8):1783-8. doi: 10.2337/dc10-0304. Epub 2010 Apr 30. PMID 20435798